CLINICAL TRIAL: NCT01126723
Title: The Effects of Tai Chi on the Nonlinear Dynamics of Frailty in Elderly Adults
Brief Title: Effects of Tai Chi on Frailty in Elderly Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-005; R37AG025037 (NIH)
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Results first posted 2015-01-30 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai Chi group (Experimental)
  Interventions: Other: Tai Chi
- Educational Control group (Active Comparator)
  Interventions: Other: Education-Control

INTERVENTIONS:
Other: Tai Chi — The Tai Chi intervention will consist of a 12 week, instructor-led, group-based Tai Chi training program (two, one-hour sessions per week).
  Arms: Tai Chi group
Other: Education-Control — The Education-Control intervention consists of a 12 week, instructor-led attention control program consisting of health education and mind-body breathing exercises (two, one-hour sessions per week)
  Arms: Educational Control group

SUMMARY:
The aim of this study is determine the effects of Tai Chi exercise, as compared to an education-based control intervention, on cardiovascular and balance system function in older people at risk of developing frailty. We hypothesize that long-term Tai Chi training will improve specific nonlinear properties associated of cardiovascular and balance dynamics in this population.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over age 70 will be included if they are able to stand and walk unassisted, are free of any acute or unstable medical conditions, and are able to understand directions and participate in the protocol.

Exclusion Criteria:

* Potential subjects will be excluded 1) if they cannot stand and ambulate unassisted, 2) are experiencing any symptomatic cardiovascular or respiratory disease, or have 3) a myocardial infarction or stroke within 6 months, 4) painful arthritis, spinal stenosis, amputation, painful foot lesions, or neuropathy that limits balance and mobility, 5) systolic BP above 160 or diastolic BP above 100 mm Hg, 6) a cardiac pacemaker, 7) Parkinson's Disease or other neuromuscular disorder, 8) metastatic cancer or immunosuppressive therapy, or 9) have significant visual impairment.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Lipsitz, MD, Principal Investigator — Hebrew Rehabilitation Center
Locations (1):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tai Chi Group | Educational Control Group
Started | 35 | 31
Completed | 29 | 28
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tai Chi Group | Educational Control Group | Total
Number analyzed (Participants) | 35 | 31 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 87 (5) | 86 (6) | 87 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 28 | 24 | 52
Frailty Index [Number; unit: participants]
  Frail | 10 | 6 | 16
  Prefrail | 20 | 23 | 43
  Nonfrail | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Frailty Index
Description: Frailty is defined as the combination of unintentional weight loss, exhaustion, low physical activity, slow walking speed, and muscular weakness.
Time Frame: post-intervention
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Tai Chi Group | Educational Control Group
Number analyzed (Participants) | 29 | 28
participants
  Frail | 7 | 5
  Prefrail | 16 | 21
  Nonfrail | 6 | 2
Statistical Analysis 1: Comparison: Tai Chi Group vs Educational Control Group; Test type: Superiority or Other; p = 0.15, Fisher Exact — The a priori threshold for statistical significance was set to 0.05

ADVERSE EVENTS:
Arm/Group | Tai Chi Group | Educational Control Group
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/31
Other Adverse Events (participants affected / at risk) | 0/35 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No